CLINICAL TRIAL: NCT07072117
Title: Comparison Between Intranasal Dexmedetomidine, Ketamine or Midazolam for Reducing Anxiety and Respiratory Complications in Children Undergoing Adenotonsillectomy
Brief Title: Intranasal Dexmedetomidine, Ketamine or Midazolam for Anxiety and Respiratory Complications in Children
Acronym: INPERM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Amira Saieed Elsayed Mousa, Dr., Zagazig University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: zagu2025-INSI; ZU-IRB#10231/11-1-2023 (Other: Zagazig University Institutional Review Board)
Record Dates: First submitted 2025-05-22; First posted 2025-07-18 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Adenotonsillectomy
Keywords: Pediatric anesthesia; Intranasal premedication; Dexmedetomidine intranasal; Ketamine intranasal; Midazolam intranasal; Preoperative anxiety; Respiratory complications; Laryngospasm in children

STUDY DESIGN:
Intervention Model Description: prospective randomized controlled clinical trial
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: The study is double-blinded. The patients and anesthesia assistant (the person evaluating the effect of the tested drug) will not be informed about tested drug. Only the anesthesiologist (the person prescribing the tested drug) will be aware.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- control group (Placebo Comparator): Patients will receive 1 mL of 0.9% saline intranasally 30 minutes before induction of anesthesia.
  Interventions: Drug: Intranasal Dexmedetomidine as a Premedication for Prevention of Anxiety & Respiratory Complications; Drug: Intranasal Ketamine as a Premedication for Prevention of Anxiety and Respiratory Complications; Drug: Intranasal Midazolam as a Premedication for Prevention of Anxiety and Respiratory Complications
- Dexmedetomidine Group (Experimental): Patients will receive 2.0 μg/kg of intranasal dexmedetomidine, diluted in 0.9% saline to a total volume of 1 mL, 30 minutes before anesthesia induction.
  Interventions: Drug: Intranasal Dexmedetomidine as a Premedication for Prevention of Anxiety & Respiratory Complications
- Ketamine Group (Experimental): Patients will receive 2 mg/kg of intranasal ketamine (50 mg/mL), diluted with 0.9% saline to a total volume of 1 mL, administered 30 minutes prior to anesthesia induction.
  Interventions: Drug: Intranasal Ketamine as a Premedication for Prevention of Anxiety and Respiratory Complications
- Midazolam Group (Experimental): Patients will receive 0.1 mg/kg of intranasal midazolam, diluted in 0.9% saline to a final volume of 1 mL, administered 30 minutes before anesthesia induction.
  Interventions: Drug: Intranasal Midazolam as a Premedication for Prevention of Anxiety and Respiratory Complications

INTERVENTIONS:
Drug: Intranasal Dexmedetomidine as a Premedication for Prevention of Anxiety & Respiratory Complications — Intranasal Dexmedetomidine as a Premedication for Prevention of Anxiety and Respiratory Complications in Children Undergoing Adenotonsillectomy
  Other Names: Intranasal Dexmedetomidine
  Arms: Dexmedetomidine Group; control group
Drug: Intranasal Ketamine as a Premedication for Prevention of Anxiety and Respiratory Complications — Intranasal Ketamine as a Premedication for Prevention of Anxiety and Respiratory Complications in Children Undergoing Adenotonsillectomy
  Other Names: Intranasal Ketamine
  Arms: Ketamine Group; control group
Drug: Intranasal Midazolam as a Premedication for Prevention of Anxiety and Respiratory Complications — Intranasal Midazolam as a Premedication for Prevention of Anxiety and Respiratory Complications in Children Undergoing Adenotonsillectomy
  Other Names: Intranasal Midazolam
  Arms: Midazolam Group; control group

SUMMARY:
This study is being done to find out which of three medications-dexmedetomidine, ketamine, or midazolam-is best at reducing anxiety and breathing problems in children having surgery to remove their tonsils and adenoids. These medicines will be given as nose drops before anesthesia. Anxiety before surgery can cause stress and lead to problems like trouble breathing during or after surgery. The study will include 148 children aged 4 to 8 years. Each child will get one of the three medicines or a placebo (saline). Researchers will observe the children for signs of anxiety before surgery and for breathing problems, such as laryngospasm, after they wake up. The goal is to find the safest and most effective medicine to help children feel calmer and breathe safely during surgery.

DETAILED DESCRIPTION:
Preoperative anxiety and respiratory complications are common in children undergoing adenotonsillectomy. Anxiety may result in behavioral changes and is associated with more difficult inductions and poorer recovery. Respiratory complications such as laryngospasm and airway obstruction are particularly dangerous in children, and minimizing these risks is a key goal of pediatric anesthesia.

Premedication with sedative drugs may help reduce anxiety and promote a smoother induction of anesthesia. The intranasal route of drug delivery is non-invasive and well tolerated in children, offering high bioavailability and avoiding the stress of IV insertion before surgery. Three commonly used intranasal medications-dexmedetomidine, ketamine, and midazolam-each have different pharmacological profiles and potential benefits.Dexmedetomidine is a selective alpha-2 adrenergic agonist that provides sedation and anxiolysis without causing respiratory depression. Ketamine is a dissociative anesthetic that reduces pain sensitivity and maintains respiratory drive. Midazolam is a benzodiazepine that provides rapid sedation and amnesia.

This randomized controlled trial will include 148 children aged 4 to 8 years undergoing adenotonsillectomy. Children will be randomly assigned to one of four groups: intranasal dexmedetomidine, ketamine, midazolam, or saline (placebo). The study is double-blinded, and the medications will be administered 30 minutes before anesthesia induction.

The primary goal is to assess and compare the incidence and severity of post-extubation laryngospasm within 30 minutes of extubation. Secondary objectives include assessing sedation level, preoperative anxiety, distress during IV cannulation, vital signs, and discharge readiness using standardized scoring systems such as the Ramsay Sedation Score, Groningen Distress Scale, and the Modified Aldrete Score.

The results of this study aim to determine the most effective and safest intranasal sedative premedication for pediatric patients, with the goal of improving surgical experiences, reducing complications, and enhancing recovery.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria
* Parent or first-degree relative acceptance
* Children with age ranged from 4 to8
* Body mass index is equal to or greater than 5th and not more than 85th percentiles
* ASA classifications Ⅰand Ⅱ
* Both sex

Exclusion Criteria:

* History of difficult intubation or extubation, cardiac, respiratory, renal and muscle diseases beside passive smoking and allergy to the tested drugs
* History of obstructive sleep apnea (OSA).
* The presence of the upper respiratory tract infection
* The need to reoperation after tonsillectomy due to hemorrhage of more than 100ml of blood during surgery
* Surgery duration is longer than 1.5 hour.

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 148 (Actual)
Dates: Start 2023-02-20 (Actual); Primary Completion 2023-08-20 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
Measurement of the vital signs mean blood pressure | From 30 minutes pre-induction to 30 minutes post-extubation (approximately 1 hour total)
  Mean arterial pressure (MAP) measured at seven time points: baseline (before intranasal drug), 10 minutes after drug administration, at induction, 10 and 30 minutes intraoperatively, and 10 and 30 minutes postoperatively.
Measurement of the heat rate | From 30 minutes pre-induction to 30 minutes post-extubation (approximately 1 hour total)
  Heart rate measured at seven time points: baseline, 10 minutes after drug administration, at induction, 10 and 30 minutes intraoperatively, and 10 and 30 minutes postoperatively.
Measurement of respiratory | From 30 minutes pre-induction to 30 minutes post-extubation (approximately 1 hour total)
  Respiratory rate measured at seven time points: baseline, 10 minutes after drug administration, at induction, 10 and 30 minutes intraoperatively, and 10 and 30 minutes postoperatively.
Scoring the incidence and severity of post-extubation laryngospasm | First 30 minutes after extubation
  Incidence and severity of laryngospasm scored using a standardized 4-point scale during the first 30 minutes after extubation.
Assessment of the sedation level done by Ramsay sedation score | First 30 minutes post-extubation
  Assessment of the sedation level done by Ramsay sedation score will be recoded at different time intervals: preoperative baseline before administration of intranasal medication, then 10 min, just before induction and 10 min, 20 min postoperative. "Ramsay Sedation Score" is described in 1974 it divides the pts level of sedation into 6 Categories ranging from severe agitation to deep coma.
Assessment of the sedation level done by Ramsay sedation score | From baseline to 20 minutes after surgery (approximately 1 hour total)
  Sedation level assessed using Ramsay Sedation Score at five time points: preoperative baseline (before drug administration), 10 minutes after drug, immediately before induction, and at 10 and 20 minutes postoperatively. The Ramsay Sedation Score is a 6-point scale ranging from anxiety/agitation to deep unresponsiveness.
Assessment of distress associated with potentially painful event using Groningen distress scale at time of canulation. | During intravenous cannulation before anesthesia induction
  (GDS) was developed to grade distress associated with a potentially painful event. It can be used to monitor a phobic patient's experience towards a triggering stimulus. The original scale was developed at the University of Groningen in The Netherland
Time to achieve discharge readiness from PACU | From arrival at PACU until Modified Aldrete Score >9 is achieved, up to 2 hours postoperatively.
  Monitoring for presence of sedation, nausea/vomiting, or other complications. Readiness assessed using Modified Aldrete Score.

CONTACTS AND LOCATIONS:
Overall Officials: Amira Saeed Kenawy, MD, Principal Investigator — Faculty of Medicine - Zagazig University
Locations (1):
- Faculty of Medicine - Zagazig University, Zagazig, Egypt

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to ethical considerations, institutional policies, and the involvement of pediatric participants. The study does not have a formal data-sharing mechanism, and the data contain potentially sensitive health information related to children.

DOCUMENTS (1):
  • Study Protocol (2023-01-11): https://cdn.clinicaltrials.gov/large-docs/17/NCT07072117/Prot_000.pdf